CLINICAL TRIAL: NCT01333254
Title: A Randomised Controlled Trial Comparing Different Methods for Short-Term Bladder Drainage in Patients With Hip Surgery
Brief Title: A Trial of Different Methods for Bladder Drainage in Hip Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Maria Halleberg Nyman, PhD, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009-075
Record Dates: First submitted 2011-04-01; First posted 2011-04-11 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Urinary Tract Infections
Keywords: urinary tract infections; urinary catheterisation
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Indwelling urinary catheter (No Intervention): Patients in this group with hip fracture will get an indwelling catheter at arrival to the orthopaedic ward. The patients with arthrosis get the indwelling catheter in the morning at the day of surgery. In both cases the indwelling catheter is inserted after shower with skin disinfectant. The catheter system is kept close. The catheter will be removed in the morning on day 2 after surgery. The patients are bladder-scanned every four-hour until normal bladder function is recaptured. If the bladder volume exceeds 400ml and the patient is unable to urinate, the patient will be re-catheterised. The procedure of the patients in this arm is in accordance with common practice in the Orthopaedic clinic.
- Intermittent urinary catheterisation (Experimental): Patients randomised to this arm will urinate either in a toilet or in a bedpan or a diaper when needed. Bladder scan control will be performed on these patients at least every four hour. If the patient is unable to urinate and bladder scan indicates ≥ 400 ml urine in the bladder, the patient will be intermittent catheterised.
  Interventions: Procedure: Intermittent urinary catheterisation

INTERVENTIONS:
Procedure: Intermittent urinary catheterisation — Patients randomised to the I group will urinate either in a toilet or in a bedpan or a diaper when needed. Bladder scan control will be performed on these patients at least every four hour. If the patient is unable to urinate and bladder scan indicates ≥ 450 ml urine in the bladder, the patient will be intermittent catheterised.
  Arms: Intermittent urinary catheterisation

SUMMARY:
The aim of the project is to evaluate differences between intermittent and indwelling catheterisation in patients with hip surgery.

Specific objectives are to determine whether:

* frequencies of urinary tract problems in hospital and up to one year after discharge differ between patient groups treated with intermittent and indwelling catheterisation respectively.
* costs and health-effects differ between the patient groups.
* experiences of urinary catheterisation differ between the patient groups

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hip fracture surgery or hip replacement due to arthrosis
* Age 50 years and above

Exclusion Criteria:

* Patients with an indwelling catheter in situ
* Cognitive impairment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Nosocomial urinary tract infection | Urine culture will be collected at admission and before discharge from the orthopaedic ward (about 5-10 days after admission)

SECONDARY OUTCOMES:
Time to normal bladder function | Hours after surgery (participants will be followed for the duration of hospital stay, about 5-10 days)
  Normal bladder function was in this study defined as a post-micturition residual urine volume of 150ml or less.The patients will be bladder-scanned every fourth hour until normal bladder function is recaptured
Costs for material and labour related to urinary catheterisation and nosocomial UTI during the first year after hip surgery | During time in hospital and up to 1 year after discharge
  Costs will be considered for material and labour. The material costs include costs for catheters, material used when inserting catheters, material used when using the bladder scan, costs for clothes and bedding changed due to urine and diapers. Also costs for medication due to urinary problems will be registered. The labour costs included are time for urinary catheterisation, bladder scan, change of patients' clothes and bedding or diapers due to urine, consultation at the Urological department or to a general practitioner due to urinary problems and length of hospital stay.
Health effects during the first year after hip surgery | Before discharge, 4 weeks, 4 months and 1 year after discharge
  The health-effects will be evaluated by EQ5D and SF-36 at discharge, 4 weeks, 4 months and 1 year after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hälleberg Nyman, RN, MSc, Principal Investigator — Örebro University Hospital, Sweden
Locations (1):
- Dept of Orthopaedic Surgery at Örebro University Hospital, Örebro, Sweden